CLINICAL TRIAL: NCT01596244
Title: Pilot and Expansion Project for the Jordan Diabetes Microclinic Project
Brief Title: Jordan Diabetes Microclinic Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microclinic International (Other)
Collaborators: Ministry of Health Jordan (Other Government); Royal Health Awareness Society (RHAS), Jordan (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WDF07-231; LT07-135 (Other Grant/Funding Number: International Diabetes Federation)
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes Mellitus, Type II
Keywords: Diabetes Mellitus, Type II; Disease management; Chronic disease; Prevention and control; Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Microclinics training (Experimental): Diabetic, pre-diabetic, or those with family members who are diabetic/pre-diabetic who participated in a 4 month long intervention with a focus on disease management, health behavior change, and social network supports in order to improve chronic disease risk factors.
  Interventions: Behavioral: Microclinic

INTERVENTIONS:
Behavioral: Microclinic — Microclinics consist of 2-8 individuals from pre-existing social networks (friends, relatives, coworkers, neighbors, etc) that voluntarily participate in ongoing education and medical monitoring from local health care professionals, learning and practicing diabetes management strategies, sharing much-needed medical supplies, and exchanging social support in the form of regular microclinic meetings.

SUMMARY:
The purpose of the study is to provide participants in economically depressed areas of Jordan essential knowledge, practical skills, and intimate support groups-called microclinics-for managing their diabetes. Microclinics consist of 2-8 individuals from pre-existing social networks (friends, relatives, coworkers, neighbors, etc) that voluntarily participate in ongoing education and medical monitoring from local health care professionals, learning and practicing diabetes management strategies, sharing much-needed medical supplies, and exchanging social support in the form of regular micro-clinic meetings.

DETAILED DESCRIPTION:
The Global Microclinic Project seeks to empower people to prevent and manage diseases in economically depressed areas Jordan. The project seeks to more broadly link health education opportunities in the form of lectures and seminars with practical experience through workshops and hands-on learning, ultimately resulting in the creation of microclinics. Microclinics are intimate support groups of diabetic patients (2-8 per clinic) who meet in their homes and businesses in order to share the costs of maintaining medical monitoring equipment and supplies, come together to support one another in the management of diabetes, collectively utilize vital treatment options, and receive personalized screening, education and management tools from medical professionals.

The microclinics concept is ideal for the management of chronic disorders such as diabetes, a disease which requires ongoing education about diet and exercise and regular monitoring of health indices such as blood glucose levels and weight change. Indeed, the microclinics model has been established successfully in the West Bank specifically to combat diabetes. The goal here is to extend the model to Jordan and to establish microclinics in a collaborative effort with the Royal Health Awareness Society (RHAS) and the Jordanian Ministry of Health (MoH).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Mentally competent
* Have diabetes or pre-diabetes or brought a family member who was diabetic/pre-diabetic (Diabetes: Fasting blood glucose higher than 125 mg/dl; Pre-diabetes: Fasting blood glucose between 100 and 124 mg/dl.)

Exclusion Criteria:

* They do not meet the above criteria
* They are pregnant
* They have significant medical complications that prevent them from making changes to diet or level of physical activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2400 (Actual)
Dates: Start 2008-04; Primary Completion 2011-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Weight (kg) | Baseline, 4 months (intervention), and 12 months (post-intervention)
  Change in weight overtime

SECONDARY OUTCOMES:
Fasting Blood Glucose (mg/dl) | Baseline, 4 months, 12 months
  Change in fasting blood glucose overtime
Hemoglobin A1c (%, HBA1c) | Baseline, 4 months, 12 months
  Change in HBA1c overtime
Body Mass Index (kg/m2) | Baseline, 4 months, 12 months
  Change in body mass index overtime

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Zoughbie, DPhil, Principal Investigator — Microclinic International; Eric Ding, PhD, Principal Investigator — Harvard University
Locations (2):
- Jordan (2):
  - Ein El-Basha Ministry of Health Center, Amman
  - Jabl Nasr Ministry of Health Center, Amman

REFERENCES:
- [Derived] Zoughbie DE, Ng TLJ, Thompson JY, Watson KT, Farraj R, Ding EL. Ramadan fasting and weight change trajectories: Time-varying association of weight during and after Ramadan in low-income and refugee populations. PLOS Glob Public Health. 2022 Oct 26;2(10):e0000371. doi: 10.1371/journal.pgph.0000371. eCollection 2022. PMID 36962504
- See also: Related Info — http://www.microclinics.org/